CLINICAL TRIAL: NCT04276311
Title: Efficacy of Rotational Atherectomy System Associated With Drug Coated Balloon Angioplasty (With or Without Stent Placement) in the Management of Lower Limb Ischemia (ELLIPSE): "Real Life" Observational Study
Brief Title: Efficacy of Rotational Atherectomy System Associated With Drug Coated Balloon Angioplasty in Limb Ischemia
Acronym: ELLIPSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSJ/02/2019
Record Dates: First submitted 2020-02-03; First posted 2020-02-19 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- symptomatic patients with complex de novo FP arterial lesions (Experimental): in symptomatic patients with claudication (Rutherford 2 and 3) and with complex de novo FP arterial lesions (TASC C).
  Interventions: Device: Percutaneous transluminal angioplasty

INTERVENTIONS:
Device: Percutaneous transluminal angioplasty — The purpose of this study is to evaluate the efficacy and the feasibility of atherectomy, using the Jetstream™ artery preparation associated to DCB treatment (Ranger™ Paclitaxel-Coated balloon), in symptomatic patients with claudication (Rutherford 2 and 3) and with complex de novo femoropopliteal arterial lesions (TASC C).

SUMMARY:
Lower extremity peripheral artery disease (PAD) is a major health problem leading to significant morbidity and even mortality. Patients with superficial femoral artery stenosis make up an important proportion of patients with PAD, and since this type of involvement was reported to be most commonly associated with intermittent claudication, this patient population has been subject to intensive research on methods to prevent disease progression and further complications.

Endovascular treatment has become the first-line treatment for low-complexity femoropopliteal (FP) lesions classified as TASC (Trans Atlantic Inter-Societal Consensus) A and B. Conversely, in case of more extensive lesions (TASC C), this treatment is still under debate because of a primary permeability that is difficult to maintain over time. Recently, studies have shown the interest of drug eluting technologies in the treatment of TASC A & B femoral-popliteal lesions, by significantly improving patency rates compared to uncoated balloons or stents.

In this context, the endovascular treatment of FP complex lesions (TASC C) continues to develop widely.

During endovascular treatment, the quality of the artery preparation has recently been identified as a factor improving outcomes. The dilatation of the artery with an uncoated balloon or POBA (Plain Old Balloon Angioplasty) is the reference method performed before stent placement or drug-coated balloons. However, some new alternatives to prepare the artery have emerged, using no more dilatation but atherectomy (Jetstream™ system).

Atherectomy appears to reduce the risk of dissections and bailout stenting and improve the acute procedural results. Its long term outcome, when associated with drug coated balloons (DCB), has recently been demonstrated in the USA to be superior to angioplasty in a single center study JET-SCE.

The purpose of this study is to evaluate the efficacy and the feasibility of atherectomy, using the Jetstream™ artery preparation associated to DCB treatment (Ranger™ Paclitaxel-Coated balloon), in symptomatic patients with claudication (Rutherford 2 and 3) and with complex de novo FP arterial lesions (TASC C).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with moderate to severe claudication: chronic symptomatic AOMI (Rutherford 2 and 3)
* Diagnosed with de novo obstructive lesions calcified in the superficial femoral artery or in P1: tight stenosis (> 70%), calcified, layered, length ˃ 10 cm or short calcified occlusions <5 cm from the superior femoral artery and P1.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.
* Affiliated to social safety plan of beneficiary under such a plan

Exclusion Criteria:

* Intra stent re-stenosis
* Recent occlusions, less than 1 month old of SFA and / or P1 (probable thrombus)
* SFA occlusion, P1 > 5 cm, from origin of SFA.
* SFA stenosis <10 cm
* Non calcified stenosis
* Participants who have participated in another research study involving an investigational product in the past 12 weeks
* Participant issuing with a safeguard measure of justice (in accordance with the low article L1122-2 of the public health code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Freedom of Target lesion revascularization | 12 months
  Percent of patients with freedom of any percutaneous intervention or surgical bypass on target lesions, performed because of restenosis or any other complication involving the target lesion

SECONDARY OUTCOMES:
Primary patency | Baseline, Month 2, Month 6, Month12, Month 24
  exempt from restenosis of the target lesion during follow-up (Doppler ultrasound)
Primary assisted patency | Baseline, Month 2, Month 6, Month12, Month 24
  patency of the target lesion following endovascular reintervention at the target vessel site in case of symptomatic restenosis (Doppler ultrasound)
Secondary patency | Baseline, Month 2, Month 6, Month12, Month 24
  patency of the target lesion after treatment of a (re)occlusion of the index lesion
Late Lumen Loss | Baseline, Month 2-Month 6
  defined as the difference between the minimal luminal diameter at the end of the procedure and the minimal luminal diameter at follow-up measured by CT Angiography.
technical success of the procedure | Day 0
  ability to pass through (intra-luminal passage) and dilate the lesion to obtain residual stenosis under angiography ≤30%.
Procedural success | Day 1
  technical success without undesirable major event observed within 24 hours post-procedure.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hopital Prive de Provence, Aix-en-Provence
  - Clinique Rhône Durance, Avignon
  - Polyclinique Notre Dame, Draguignan
  - Hopital Europeen, Marseille
  - Hôpital Saint Joseph, Marseille
  - Clinique Saint Georges, Nice
  - Clinique Les Franciscaines, Nîmes
  - Polyclinique Les Fleurs, Ollioules

IPD SHARING:
Plan to Share IPD: No